CLINICAL TRIAL: NCT03747016
Title: The Use of High-energy Digestible Food in Women Undergoing Caesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ERAS obstetric
Record Dates: First submitted 2018-11-04; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Caesarean Section
MeSH Terms: interventions — methyl N-acetylsibirosaminide

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- High energy 2 (Experimental): In the second step, the experimental group (Group E2) was given high energy digestible food 300ml before the time of gastric emptying found in the first step before surgery.
  Interventions: Dietary Supplement: high-energy digestible food E2
- Glucose 2 (Active Comparator): In the second step, Group G2 is given 5% glucose injection 300ml before the time of gastric emptying found in the first step before surgery.
  Interventions: Dietary Supplement: glucose injection G2
- Normal saline 2 (Placebo Comparator): In the second step, Group N2 is given normal saline 300ml before the time of gastric emptying found in the first step before surgery.
  Interventions: Dietary Supplement: normal saline N2
- Control 2 (No Intervention): In the second step, the control group (Group C2) was not given any diet before surgery.
- High energy 1 (Experimental): In the first step,The experimental group (Group E1) is treated with high energy digestible food 300ml.
  Interventions: Dietary Supplement: high-energy digestible food E1
- Glucose1 (Active Comparator): In the first step, Group G1 is given 5% glucose injection 300ml
  Interventions: Dietary Supplement: glucose injection G1
- Normal saline 1 (Placebo Comparator): In the first step, Group N1 is given normal saline 300ml.
  Interventions: Dietary Supplement: normal saline N1

INTERVENTIONS:
Dietary Supplement: high-energy digestible food E2 — The women undergoing Cesarean section are given high energy digestible food 300ml before surgery
  Other Names: E2
  Arms: High energy 2
Dietary Supplement: glucose injection G2 — The women undergoing Cesarean section are given glucose injection 300ml before surgery
  Other Names: G2
  Arms: Glucose 2
Dietary Supplement: normal saline N2 — The women undergoing Cesarean section are given normal saline 300ml before surgery
  Other Names: N2
  Arms: Normal saline 2
Dietary Supplement: high-energy digestible food E1 — The women in delivery room are given high energy digestible food 300ml.
  Other Names: E1
  Arms: High energy 1
Dietary Supplement: glucose injection G1 — The women in delivery room are given glucose injection 300ml.
  Other Names: G1
  Arms: Glucose1
Dietary Supplement: normal saline N1 — The women in delivery room are given normal saline 300ml.
  Other Names: N1
  Arms: Normal saline 1

SUMMARY:
Traditionally, Fasting for more than 8 hours before operation is administered to reduce the risk of reverse flow and aspiration. ASA guidelines suggest a 2-hour fasting for clear fluid in healthy people before elective surgery. But in delivery women, the gastric emptying time is affected by the physiological change. This study is a prospective randomized controlled study to investigate the gastric emptying time of high energy digestible foods in delivery women, and the effect of high energy digestible food given before surgery on the comfort and metabolism of women undergoing Cesarean section. In the first step, 60 women in delivery room whose gastric volume less than 3.81 cm2 are randomly divided into three groups, 20 cases in each group. The experimental group (Group E1) is treated with high energy digestible food 300ml, Group G1 is given 5% glucose injection 300ml and Group N1 is given normal saline 300ml. The gastric volume was determined by ultrasonography once every hour until gastric volume less than 3.81cm2, and the time of gastric emptying was determined. The second step was to recruit 80 cases of full-term elective cesarean section. They were randomly divided into four groups, 20 cases in each group. The experimental group (Group E2) was given high energy digestible food 300ml before the time of gastric emptying found in the first step , Group G2 is given 5% glucose injection 300ml and Group N2 is given normal saline 300ml, while the control group (Group C2) was not given any diet. After admission to the operation room, the volume of the stomach was measured by ultrasound, and the differences of comfort, body temperature, shivering, blood glucose and postoperative anal exhaust time between the two groups were observed. This study is going to investigate the gastric emptying time of high energy digestible foods in delivery women, and the effect of high energy digestible food on the comfort, body temperature and blood glucose of women undergoing Cesarean section, so as to provide a good basis for reducing the surgery stress in women undergoing Cesarean section.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled study to investigate the gastric emptying time of high energy digestible foods in delivery women, and the effect of high energy digestible food given before surgery on the comfort and metabolism of women undergoing Cesarean section.

In the first step, 60 women in delivery room are enrolled, who are full term singleton pregnancy subjects ranging 18 to 50 years old and fasting for more than 8 hours. They are randomly divided into three groups, 20 cases in each group.

The experimental group (Group E1) is treated with high energy digestible food 300ml, Group G1 is given 5% glucose injection 300ml and Group N1 is given normal saline 300ml. The gastric volume was determined by gastric antrum cross-sectional area (CSA) measured with ultrasonography before drinking and once every hour after drinking. Once CSA is less than 3.81 cm2, the time is recorded as gastric emptying time of the woman. The overall gastric emptying time of high energy digestible food is determined with the 90 percentile gastric emptying time of women drinking high energy digestible food.

The second step was to recruit 80 cases of full-term elective cesarean section. They were randomly divided into four groups, 20 cases in each group. The experimental group (Group E2) was given high energy digestible food 300ml before the time of gastric emptying found in the first step, Group G2 is given 5% glucose injection 300ml and Group N2 is given normal saline 300ml, while the control group (Group C2) was not given any diet. After admission to the operation room, the volume of the stomach was measured by ultrasound, and the differences of comfort, body temperature, shivering, blood glucose and postoperative anal exhaust time between the two groups were observed.

This study is going to investigate the gastric emptying time of high energy digestible foods in delivery women, and the effect of high energy digestible food on the comfort, body temperature and blood glucose of women undergoing Cesarean section, so as to provide a good basis for reducing the surgery stress in women undergoing Cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologist) grade II, full term singleton pregnancy subjects aged 18 to 50 years old;
* subjects undergoing elective cesarean section under combined spinal epidural anesthesia;
* volunteered to participate in the study and signed informed consent.

Exclusion Criteria:

* related drug allergies or taboo;
* Severe cardiopulmonary disorders (New York Heart Association Classification III-IV, or left ventricular ejection fraction < 30%) and liver and kidney dysfunction (alanine aminotransferase exceeding the upper limit of normal value twice, creatinine exceeding the upper limit of normal value 1.5 times), alcoholism history;
* there are metabolic diseases such as gestational diabetes mellitus, or using drugs that affect metabolism;
* the subjects were unable to cooperate or to communicate;
* the subjects suffered from psychosocial diseases;
* participated in other clinical trials within one month;
* there is drug abuse.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
body temperature | the time point when newborn delivers and 1 hour after surgery
  Maternal tympanic temperature measured by infrared ear thermometer

SECONDARY OUTCOMES:
Maternal comfort | up to 24 hours after surgery
  Maternal comfort is measured by the women undergoing Cesarean section with visual analogy scale. Respondents mark the location on the 10-centimeter line corresponding to the amount of comfort they experienced.
Incidence and severity of shivering | up to 1 hour after surgery
  Incidence and severity of shivering is assessed with Wrench's Grade.
nausea and vomitting after surgery | up to 24 hours after surgery
  The severity of postoperative nausea and vomitting is assessed with CTCAE v4.0.
flatus time | up to 48 hours after surgery
  The time point when anal exhaust restarts after surgery
pain after surgery | up to 48 hours after surgery
  Maternal pain is measured by the women undergoing Cesarean section with visual analogy scale. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain they experienced.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First Maternity and Infant Hospital, affiliated to Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided